CLINICAL TRIAL: NCT02552797
Title: The Development and Piloting of 'Power Up': a Tool for Young People with Internalising/emotional Disorders to Make Shared Decisions in Child and Adolescent Mental Health Services (CAMHS)
Acronym: Power Up
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Changes to scope of project and funding
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 15/0340
Record Dates: First submitted 2015-08-27; First posted 2015-09-17 (Estimated); Last update posted 2024-12-04 (Actual); Status verified 2015-09

CONDITIONS: Internalising Disorders; Anxiety; Depression
Keywords: Shared Decision Making; CAMHS
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Using Power Up (Experimental): Participants will use 'Power Up' to help them make shared decisions about their treatment or care
  Interventions: Behavioral: Shared Decision Making tool
- Not using Power Up (No Intervention): Participants will continue treatment as usual

INTERVENTIONS:
Behavioral: Shared Decision Making tool
  Arms: Using Power Up

SUMMARY:
Patients should be able to have a say in their care and treatment, but how this should work for children and young people with mental health difficulties is unknown. For example, how and when do young people want to be involved in decision making, and what is important to them, their parents/guardians and healthcare professionals? This project will address these questions and will develop a tool known as 'Power Up' to help young people with mental health difficulties make decisions about their own care and treatment.

This project will run for 24 months and will:

1. Understand the beliefs, experiences, and values of young people, their parents/guardians and clinicians around shared decision making (SDM) in mental health.
2. Use these responses to develop 'Power Up'; a tool to help young people make decisions about their care or treatment in mental health services.
3. Pilot 'Power 'Up' in child and adolescent mental health services to estimate the number of patients who would want to use Power Up and to see whether patients can be recruited and followed up with measures. The pilot study would investigate randomisation, see how clinicians cooperate, and identify barriers to collaboration and ways of overcoming these.

Forty five young people, parents and clinicians will be recruited for interviews and focus groups to inform tool development. Sixty young people aged 1116 will be recruited for the pilot/feasibility study. Measurements will be collected at baseline, session by session, and at the end of treatment.

DETAILED DESCRIPTION:
TOOL DEVELOPMENT All potential information about the project can be given verbally (this will be over the phone in the first instance). For CYP (children and young people) that are under 16, parental consent will also be needed. After the phone call, if individuals are interested in taking part, age appropriate information sheets will be posted out to both the CYP and guardians/parents outlining the details of the study. The researcher will discuss any questions potential participants may have over the telephone, and both will have as long as they need to decide whether to take part. If they decide to take part the participants will be invited to take part if they meet study inclusion criteria. For clinicians, the researcher will come to staff meetings, outline the study and leave contact details/expression of interest forms so that those who are interested can get in contact to find out more. For young people and families, clinician's will briefly outline the study and interested participants will fill out an expression of interest form. After the researcher receives the contact details participants will be contacted by a researcher so that further information researcher will then arrange a time to meet with them for an interview or when they may be available for a focus group, and consent forms will be signed. Clinicians, parents/guardians and those aged 16 will also have the opportunity to have the interview conducted over the phone if they prefer (in which case consent forms will be posted). During interviews participants will speak about their previous experiences and beliefs about SDM as well as view and discuss the few existing SDM tools used with young people within CAMHS to use as a baseline for further development. After the interview participants will be debriefed, and be given the opportunity to validate themes that emerge from the data once analysed.

USING POWER UP IN CAMHS SERVICES Clinicians For clinicians, the researcher will be come to staff meetings, outline the study and leave contact details/expression of interest forms so that those who are interested can get in contact to find out more. After the researcher receives the clinicians contact details they will be contacted by a researcher so that further information about the project can be given verbally (this will be over the phone in the first instance). The researcher will then meet with those who are interested an outline the study to them (including randomisation). The researcher will discuss any questions potential participants may have over the telephone, and both will have as long as they need to decide whether to take part. Those who want to take part will be asked to sign a consent form, and will be allocated to use 'Power Up' or continue as TAU with their patients.

CYP/ Families Young people and their families will be invited to take part if they meet the study criteria. Clinicians will briefly outline the study and interested participants will fill out an expression of interest form. After the researcher receives the contact details patients and their families will be contacted by a researcher so that further information about the project can be given verbally (this will be over the phone in the first instance). For CYP's that are under 16, parental consent will also be needed. After the phone call, if individuals are interested in taking part, age appropriate information sheets will be posted out to both the CYP and Guardians/Parents outlining the details of the study. The researcher will discuss any questions potential participants may have over the telephone, and both will have as long as they need to decide whether to take part.

If they decide to take part the researcher will then arrange a time to meet with them at the CAMHS service and complete any baseline assessments (week 1) for clinical symptomology (e.g. Revised Child Anxiety and Depression Scale , Strengths and Difficulties Questionnaire) if these are not routinely collected by the CAMHS service. Randomisation will occur at clinician level and participants will be made aware of this in the information sheets. Throughout the course of treatment session by session measures at weeks 2, 4 and 8) will be completed. Participants and clinicians will also be asked if they consent to the researcher observing one appointment session when the tool is being used (this is optional and will last up to 30 mins, but will likely be week 2 or 3) to understand how the tool is being used in clinical settings.

At the end of treatment (approximately week 8) clinical symptomology, therapeutic alliance, level of shared decision making, and experience of care will be collected. Participants will be invited for an interview to hear their views and experiences about the 'Power Up tool' which like other interviews will take place at a time of their choosing and abide by SOPs (standard operating procedures). Participants will exit the trial and any further treatment will be discussed between them and their healthcare professional.

ELIGIBILITY:
Inclusion Criteria:

1. A young person between 11 and 16 years of age with an emotional/internalising disorder who is accessing CAMHS.
2. A parent/guardian of a young person between 11 and 16 years of age with an emotional/internalising disorder who is accessing CAMHS.
3. A clinician in a participating CAMHS site.
4. Only those providing consent will be included. Where potential participants are under 16 parents/legal guardians will also have to provide consent.

Exclusion Criteria:

1. Any individual who is not accessing a participating CAMHS site.
2. Given there are no additional resources for an interpreter, children or parents who are not comfortable with English may not be included
3. Young people under the age of 11, or over the age of 16 would not be included.
4. Parents/guardians of young people with SEN (special educational needs) will not be included
5. Those who do not consent.

Min Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Shared Decision Making Questionnaire (CollaboRATE) | Level of Shared Decision Making at end of treatment (this will be at approximately week 8)
  A measure of SDM - this consists of three questions related to shared decision making on a 9 point likert scale ranging from 0 'no effort was made' to 9 'every effort was made'.

CONTACTS AND LOCATIONS:
Overall Officials: Julian Edbrooke-Childs, PhD, Principal Investigator — University College London and Anna Freud Centre

REFERENCES:
- [Derived] Edbrooke-Childs J, Edridge C, Averill P, Delane L, Hollis C, Craven MP, Martin K, Feltham A, Jeremy G, Deighton J, Wolpert M. A Feasibility Trial of Power Up: Smartphone App to Support Patient Activation and Shared Decision Making for Mental Health in Young People. JMIR Mhealth Uhealth. 2019 Jun 4;7(6):e11677. doi: 10.2196/11677. PMID 31165709